CLINICAL TRIAL: NCT02714933
Title: Thoracic Imaging in Children With Neither Irradiation Nor Injection, by a New MRI Protocol Including Advanced Zero Time Echo (ZTE)
Brief Title: Thoracic MRI Imaging in Children
Acronym: ImagINI-CHEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P150909; 2016-A00416-45 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease
Keywords: pulmonary; parenchyma; MRI sequence Advanced ZTE; chest computed tomography
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI sequence Advanced ZTE (Experimental)
  Interventions: Other: MRI sequence Advanced ZTE

INTERVENTIONS:
Other: MRI sequence Advanced ZTE — Evaluation of the image quality in terms of visualization of anatomical structures of the lung parenchyma in safe zone by a new imaging method of the pulmonary parenchyma by MRI (Advanced ZTE sequence).

SUMMARY:
The aim of this study is to compare a new Magnetic Resonance Imaging (MRI)protocol, including a new MRI sequence for visualization of lung parenchyma, to computed tomography as the gold standard for the evaluation of thoracic region in children.

DETAILED DESCRIPTION:
The potential effects of ionizing radiation are of particular concern in children. Exposure to ionizing radiation of medical origin is responsible for an increased risk of brain tumors and hematopoietic lineage in children. It is therefore necessary to find alternative to the use of irradiating imaging examinations. Currently, computed tomography (CT) is the gold standard in the study of lung diseases and is used in children deepening of standard radiography in acute or chronic situations, sometimes requiring iterative controls. Chest CT delivers a radiation dose equivalent to up to 500 days of natural exposure. Moreover, for the analysis of mediastinal and vascular structures it requires an intravenous injection of iodinated contrast, potentially source of nephrotoxicity and anaphylactic reactions. Recently, new developments in Magnetic Resonance Imaging (MRI) have shown interest in the study of lung diseases when they are responsible for filling of aeric structures (mucoid impaction in cystic fibrosis, alveolar filling in infectious process and tumor) and in the analysis of vascular and mediastinal structures and heart. However, the aerated lung presenting a very low density of protons, and MRI being particularly sensitive to artifacts from cardiac and respiratory movements, sequences currently used in MRI remain insufficient in the analysis of pulmonary structures and pathologic conditions not filling aeric spaces (bronchial, cystic, emphysematous or interstitial diseases). The aim of this study is to test in clinical practice, a new MRI sequence for visualizing lung parenchyma, 3D zero Time Echo (Advanced ZTE) and to propose a protocol combining several MRI sequences without injection as an alternative to chest CT with or without contrast medium injection in childhood.

The proposed hypotheses are :

1. MRI sequence Advanced ZTE allows visualization of normal and pathological lung parenchymal structures.
2. A complete MRI protocol, without injection, including this sequence to those already used in clinical practice could replace the enhanced CT in most pediatric indications.

The principal objective of the study is to evaluate the Advanced ZTE sequence in the visualization of lung parenchyma structures in comparison to CT scan in lung window as gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 6-16 years,
* Introducing one or more clinical indications for performing a chest CT with and without contrast injection within 1 day to 3 months.
* Monitoring at the Necker Hospital.
* Signature of consent by a holder of parental authority.
* Patient affiliated or beneficiary of a social security

Exclusion Criteria:

* Contraindication to performing MRI: claustrophobia, cochlear implant, nerve stimulator, pacemaker implant or intra-cardiac metallic foreign body, chest or eye.
* Need for MRI under sedation or general anesthesia.
* Indication of an emergency CT within less than 12 hours (especially suspected pulmonary embolism).

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Score on the Likert Scale of visual image quality | 3 months
  Evaluation MRI sequence Advanced ZTE in terms of image quality and visualization of the pulmonary parenchyma

SECONDARY OUTCOMES:
Noise index | 3 months
  Quantitative evaluation for the quality of the image obtained by the Advanced ZTE sequence
Contrast index | 3 months
  Quantitative evaluation for the quality of the image obtained by the Advanced ZTE sequence
visual score of image quality in CT in parenchyma window in safe area | 3 months
visual score of image quality in CT in pulmonary parenchyma lesions | 3 months
visual score of image quality in MRI in parenchyma window in safe area | 3 months
visual score of image quality in MRI in pulmonary parenchyma lesions | 3 months
visual score of image quality in CT viewing the normal structures of the mediastinum | 3 months
visual score of image quality in CT viewing the mediastinal and pleural lesions or abnormalities | 3 months
visual score of image quality in MRI viewing the normal structures of the mediastinum | 3 months
visual score of image quality in MRI viewing the mediastinal and pleural lesions or abnormalities | 3 months
Number of participants with adverse events in CT | 3 months
Number of participants with adverse events in MRI | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: laureline BERTELOOT, MD, PhD, Principal Investigator — Hopital Necker, Assitance Publique-Hôpitaux de Paris
Locations (1):
- Necker hospital, Paris, paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drummond D, Marquant F, Zanelli E, Lozach C, Boddaert N, Taam RA, Neven B, Le Bourgeois M, Hadchouel A, Sarnacki S, Elie C, Delacourt C, Berteloot L. Radiation-free and injection-free imaging of the paediatric chest using a magnetic resonance imaging protocol including zero time echo sequence (3D-ZTE). Eur J Pediatr. 2024 Oct;183(10):4297-4308. doi: 10.1007/s00431-024-05678-1. Epub 2024 Jul 27. PMID 39066822
- [Background] Gorkem SB, Coskun A, Yikilmaz A, Zurakowski D, Mulkern RV, Lee EY. Evaluation of pediatric thoracic disorders: comparison of unenhanced fast-imaging-sequence 1.5-T MRI and contrast-enhanced MDCT. AJR Am J Roentgenol. 2013 Jun;200(6):1352-7. doi: 10.2214/AJR.12.9502. PMID 23701075
- [Background] Liszewski MC, Hersman FW, Altes TA, Ohno Y, Ciet P, Warfield SK, Lee EY. Magnetic resonance imaging of pediatric lung parenchyma, airways, vasculature, ventilation, and perfusion: state of the art. Radiol Clin North Am. 2013 Jul;51(4):555-82. doi: 10.1016/j.rcl.2013.04.004. PMID 23830786
- [Background] Johnson KM, Fain SB, Schiebler ML, Nagle S. Optimized 3D ultrashort echo time pulmonary MRI. Magn Reson Med. 2013 Nov;70(5):1241-50. doi: 10.1002/mrm.24570. Epub 2012 Dec 4. PMID 23213020